CLINICAL TRIAL: NCT02203799
Title: Immune Responses in Peanut Allergic Subjects Undergoing Peanut Oral Immunotherapy
Brief Title: Peanut Oral Immunotherapy in Children With Peanut Allergy (Peanut Flour)
Acronym: PeanutFlour
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Carla McGuire Davis, Associate Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 26819
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2024-01-19 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2023-04

CONDITIONS: Peanut Allergic Subjects
Keywords: Peanut Allergy; Anaphylaxis; Desensitization; Food Allergy; Oral Immunotherapy
MeSH Terms: conditions — Peanut Hypersensitivity; Anaphylaxis; Food Hypersensitivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Peanut Oral Immunotherapy (POIT) (Experimental): The peanut OIT is taken in the form of peanut flour. It will be given in small cups containing the amount of flour that needs to be eaten for one dose. One dose should be taken per day.
  Interventions: Biological: Peanut Oral Immunotherapy (POIT)

INTERVENTIONS:
Biological: Peanut Oral Immunotherapy (POIT) — The peanut protein is ingested in the form of peanut flour. Peanut flour will be given in small pre-measured soufflé cups containing the amount of peanut flour that needs to be eaten for one dose. One dose will be taken per day. Dosage of the peanut flour will begin with 1.8 mg of peanut protein during the initial visit or the lowest tolerated dose on initial challenge and increased every 2 during the build-up phase until the maintenance dose of peanut protein (3900 mg) is reached.
  Other Names: Peanut Flour; Peanut Oral Immunotherapy

SUMMARY:
Many children who are allergic to peanuts do not outgrow their allergy and have very severe allergic reactions called anaphylaxis. Symptoms of anaphylaxis include difficulty breathing, decreased blood pressure, hives, and lip or throat swelling after exposure to an allergen. A severe allergic reaction can lead to death if not treated appropriately.

The purpose of this study is to find out if there is a way to treat children with peanut allergy to help lower the risk of severe allergic reactions and also cause them to lose their allergy to peanuts. The approach that will used for this study is a process called "desensitization".

Oral immunotherapy involves eating gradually increasing amounts of a food over several months. This is a research study because at this time peanut oral immunotherapy (OIT) is investigational. Peanut OIT (study drug) is investigational because it is not currently approved for clinical use by the Food and Drug Administration. There are no alternative safe and effective treatments for peanut induced allergic reactions other than peanut avoidance and treatment with medications.

DETAILED DESCRIPTION:
This is a phase I, open label study for the initial 12 month desensitization phase of peanut oral immunotherapy and a 2 year maintenance phase. Subjects will be recruited to determine the immune response during the administration of peanut OIT after the development of disease. Cohort will include children age 5-16 years who have peanut allergy. The study will require approximately 36 visits with 3 phases: screening phase (~ 2 months); build-up phase (weeks 1 year), followed by the maintenance phase (2 years).

The primary objective of the OIT protocol is to desensitize subjects to peanut and this occurs over the first 12 months of the study (build-up phase). The first dose will be based on the amount at which the subject reacted during a double blind placebo controlled food challenge (DBPCFC). Thereafter, dose escalation would continue as outlined in the protocol for approximately 50 weeks until the maintenance dose of peanut protein (3900 mg) is reached.

The maintenance phase will continue from the end of the build-up phase until approximately 24 months. During this phase, the subject will switch to a peanut equivalent dose for the maintenance phase. At the conclusion of the maintenance phase a DBPCFC will be done. Negative challenges will be confirmed by open challenge. DBPCFC will be done.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-16 years of either sex, any race, any ethnicity, weighing at least 18.3 kg at the time of the initial visit.
* The presence of Immunoglobulin E (IgE) specific to peanuts (a positive skin prick test to peanuts (diameter of wheal > 3.0 mm) and a positive in vitro IgE [CAP-FEIA] > 7 kUA/L) measured within the past year.
* Significant clinical symptoms occurring within 120 minutes after ingesting peanuts during an observed DBPCFC. Patients who have not had previous oral exposure to peanut will be observed for a longer duration of 150 minutes because they may demonstrate a delayed immune response, given the lack of prior peanut exposure. Also, patients with a history of prior anaphylaxis will be observed for 150 minutes.
* Provide signed informed consent.
* Ability to follow-up regularly for scheduled appointments.
* Subjects will not be excluded if they are primarily Spanish speaking.
* Females of childbearing potential must be willing to practice an acceptable form of birth control throughout the protocol.
* Epinephrine injection training provided. Participant has current in-date epinephrine injector and parent/guardian demonstrates proper use

Exclusion Criteria:

* History of severe anaphylaxis to peanut as defined by hypoxia, hypotension, or neurological compromise (Cyanosis or SpO2 < 92% at any stage, hypotension, confusion, collapse, loss of consciousness; or incontinence)
* Currently participating in a study using an investigational new drug.
* Participation in any interventional study for the treatment of food allergy in the past 12 months or while participating in this study.
* Poor control or persistent activation of atopic dermatitis.
* Diagnosis of persistent asthma as defined by NHLBI criteria and currently being treated with daily doses of inhaled corticosteroids or requiring a rescue inhaler more than 2 days per week.
* Inability to discontinue antihistamines for skin testing and Oral Food Challenges (OFCs).
* Pregnant female.
* Chronic medical condition requiring frequent use of oral steroids, chronic psychiatric illness or history of substance abuse.
* Active eosinophilic esophagitis requiring medication therapy during the past 12 months.
* Subjects with known oat or wheat allergy
* Subjects currently on the build-up phase of environmental allergy immunotherapy injections
* Live more than 175 miles away from Texas Children's Hospital located in the Medical Center.

Ages: 5 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2014-07-31 (Actual); Primary Completion 2020-02-11 (Actual); Study Completion 2020-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla M Davis, MD, Principal Investigator — Texas Children's Hospital/Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began on 7/31/2014 and the last subject was recruited on 12/23/2016.
  Participants were recruited from the Food Allergy Program at Texas Children's Hospital and by referral from community physicians.
Pre-assignment Details: Participants were brought in for a screening visit to assess for eligibility in the study. 28 subjects were seen for screening visit and 13 subjects were ineligible due to failure to complete food challenge (1), FEV1<90% predicted on spirometry (4), Peanut IgE < 7 kU/L (1), and were not interested due to time commitment (5), unable to tolerate initial dose (2).
Period: Overall Study
Arm/Group | Peanut Oral Immunotherapy (POIT)
Started | 15
Completed | 12
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Arm/Group | Peanut Oral Immunotherapy (POIT)
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.74 (2.42)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Number of Participants that Completed the Protocol [Count of Participants; unit: Participants] — Number of Participants that Completed the Protocol
  Participants
    Withdrawal | 3
    Completed | 12

OUTCOME MEASURES:

1. Primary Outcome: Determine the Percentage of Patients Tolerating the 12-month DBPCFC
Description: Patients underwent a build-up phase (month 0-12). The patients returned every 2 weeks during the build-up phase until the maintenance dose of 3900 mg was achieved. The 12-month double blind placebo controlled food challenge (DBPFC) was performed on achieving the maintenance dose. The primary objective was to determine the percentage of subjects tolerating a cumulative dose of 26255 mg of peanut flour with absence of clinical symptoms during the 12-month DBPCFC.
Time Frame: Month 12 after first dose of peanut flour
Population: Three (3) subjects withdrew from the trial prior to maintenance phase. Only 12 subjects were analyzed for this objective.
Measure: Count of Participants; unit: Participants
Groups:
- Percentage of Subjects Who Tolerated 6000mg: The percentage of subjects who tolerated 6000mg at the double-blind placebo control food challenge after completing the build-up phase (50 weeks). The participant was challenged to the following doses: 75, 150, 500, 1000, 2000, 3000, 4000, 4500, 5000, and 6000 mg of peanut protein. The doses were given every 15 minutes in the form of peanut flour.
Arm/Group | Percentage of Subjects Who Tolerated 6000mg
Number analyzed (Participants) | 12
Participants
  Tolerated | 2
  Did not tolerate | 10

2. Secondary Outcome: Sustained Unresponsiveness After 1 Month of Treatment Discontinuation
Description: To compare the change in dose tolerated after one month of abstaining from peanut to determine sustained unresponsiveness. The subjects underwent a DBPCFC at month 36 and month 37. The mean of the highest dose tolerated by the subjects was assessed at these two timepoints.
Time Frame: Month 36 and 37 after first dose of peanut flour
Population: Nine (9) patients did not complete the food challenge after one month of abstaining from peanut. Six (6) patients were analyzed.
Measure: Mean (Standard Error); unit: mg
Groups:
- Dose Tolerated After One Month of Abstaining: To compare the dose tolerated after one month of abstaining from peanuts to determine sustained unresponsiveness, we assessed the percentage of subjects who tolerated 6000 mg at the double-blind placebo control food challenge after completing the build-up phase. The participant was challenged to the following doses: 75, 150, 500, 1000, 2000, 3000, 4000, 4500, 5000, and 6000 mg of peanut protein. The doses were given every 15 minutes in the form of peanut flour.
Arm/Group | Dose Tolerated After One Month of Abstaining
Number analyzed (Participants) | 6
mg
  37 month challenge | 1010.88 (835.33)
  36 month challenge | 2736.67 (854.70)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the build up phase (ranged from 50-71 weeks for the eligible participants) and 2 years of the maintenance phase.
Groups:
- Frequency of Symptom Occurrence During Dosing: Frequency of Symptom Occurrence During Dosing which was as follows: 1.8, 3.6, 7.2, 14.4, 28.8, 40, 60, 80, 100, 120, 240, 300, 450, 600, 750, 900, 1050, 1200, 1350, 1500, 1800, 2100, 2400, 3000, 3600, and 3900 mg of peanut protein daily with every 2 week up-dosing. Participants maintained daily dosing of 3900 mg of peanut protein for 24 months.
Arm/Group | Frequency of Symptom Occurrence During Dosing
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 15/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Frequency of Symptom Occurrence During Dosing (N=15)
Rash (Skin and subcutaneous tissue disorders) | 13
Skin Itchiness (Skin and subcutaneous tissue disorders) | 13
Hives (Skin and subcutaneous tissue disorders) | 12
Sneezing/Itching (Respiratory, thoracic and mediastinal disorders) | 8
Stuffy Nose (Respiratory, thoracic and mediastinal disorders) | 7
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 8
Throat Symptoms (Respiratory, thoracic and mediastinal disorders) | 10
Wheezing (Respiratory, thoracic and mediastinal disorders) | 4
Gastrointestinal, Subjective Complaints (Gastrointestinal disorders) | 9
Gastrointestinal, Objective Complaints (Gastrointestinal disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/99/NCT02203799/Prot_SAP_000.pdf